CLINICAL TRIAL: NCT02563418
Title: Feasibility of a Video-oculography in Patients With Huntington's Disease VOG-HD Study
Acronym: VOG-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2013 - 11
Record Dates: First submitted 2015-09-08; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Huntington Disease
Keywords: video oculography
MeSH Terms: conditions — Huntington Disease | interventions — Eye-Tracking Technology

ARMS (1):
- Patient with Huntington's disease (Experimental)
  Interventions: Device: Eye-tracking

INTERVENTIONS:
Device: Eye-tracking

SUMMARY:
The purpose of this study is to know the limits of feasibility of a reliable oculomotor record for patient with Huntington's disease.

ELIGIBILITY:
Inclusion Criteria:

* Corrected visual acuity >1/10
* Aged over 18 years
* Patient with the mutation that is to say the presence of an abnormal number of trinuclide: CAG> 38 in the first exon of the huntingtin gene.
* Total Functional Capacity Scale (CFT) ≥ 3

Exclusion Criteria:

* Patients or trustworthy person who have not given their written consent, informed and signed.
* Patients are not affiliated or who are not entitled to Social Security
* Private patients of liberty by administrative or judicial decision, or patients supervision
* Associated disease with neurological repercussions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
saccadic measures with the eye tracker | 1 day
  one measure in the evening and one in the afternoon

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Angers, France